CLINICAL TRIAL: NCT03620266
Title: Effects of Bilberry and Oat Intake on Plasma Lipid Profile, Inflammation, and Exercise Capacity in Patients With Type 2 Diabetes and/or Myocardial Infarction (BioDiaMI): a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Effects of Bilberry and Oat Intake After Type 2 Diabetes and/or MI
Acronym: BioDiaMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ole Frobert, MD, PhD (Other)
Collaborators: Region Västmanland (Other); Region Skane (Other); Chalmers University of Technology (Other); Värmland County Council, Sweden (Other Government); Vastra Gotaland Region (Other Government); Aarhus University Hospital (Other); Odense University Hospital (Other); Falu Hospital (Other)
Responsible Party: Sponsor-Investigator, Ole Frobert, MD, PhD, Professor, Region Örebro County
Organization: Region Örebro County (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BioDiaMI
Record Dates: First submitted 2018-08-02; First posted 2018-08-08 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Myocardial Infarction
Keywords: acute myocardial infarction; diet therapy; anthocyanin; bilberry bush; exercise capacity; cholesterol; beta glucans; type 2 diabetes mellitus
MeSH Terms: conditions — Myocardial Infarction; Diabetes Mellitus, Type 2 | interventions — Vaccinium myrtillus extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Bilberry (Experimental): Dietary supplement with bilberry shakes 2 times daily for 3 months (containing in total 40g of dried bilberry powder equalling 480 g of fresh berries per day). Product development in collaboration with Glucanova AB.
  Interventions: Dietary Supplement: Bilberry
- Reference/Placebo (Placebo Comparator): Dietary supplement with reference shakes 2 times daily for 3 months (containing no active bilberry or no active oats, but with similar texture and taste as both bilberry and oat). Product development in collaboration with Glucanova AB.
  Interventions: Dietary Supplement: Placebo
- Bioprocessed oat bran (Experimental): Dietary supplement with bioprocessed oat bran shakes 2 times daily for 3 months (containing beta glucans from the Glucanova® technology, invented by Glucanova AB).Product development in collaboration with Glucanova AB.
  Interventions: Dietary Supplement: Bioprocessed oat bran
- Combination of oat and bilberry (Experimental): Dietary supplement with a combination of bioprocessed oat bran and dried bilberry (shakes) 2 times daily for 3 months. Product development in collaboration with Glucanova AB.
  Interventions: Dietary Supplement: Combination bilberry/oats

INTERVENTIONS:
Dietary Supplement: Bilberry — The dietary intervention will continued for three months. After randomization, participants will be given bilberry shakes (active), liquid oat shakes (active), a combination shake with bilberry and oats, or reference shakes (placebo product containing no active bilberry or active oats but with similar taste and texture as both oat and bilberry), for intake two times a day (t.i.d). The formula for the shakes to be used in the intervention will be finalized during the initial project period.
  Arms: Bilberry
Dietary Supplement: Placebo — The dietary intervention will be continued for three months. After randomization, participants will be given bilberry shakes (active), liquid oat shakes (active), a combination shake with bilberry and oats, or reference shakes (placebo product containing no active bilberry or active oats but with similar taste and texture), for intake two times a day (t.i.d). The formula for the shakes to be used in the intervention will be finalized during the initial project period.
  Arms: Reference/Placebo
Dietary Supplement: Bioprocessed oat bran — The dietary intervention will be continued for three months. After randomization, participants will be given bilberry shakes (active), liquid oat shakes (active), a combination shake with bilberry and oats, or reference shakes (placebo product containing no active bilberry or active oats but with similar taste and texture), for intake two times a day (t.i.d). The formula for the shakes to be used in the intervention will be finalized during the initial project period.
  Arms: Bioprocessed oat bran
Dietary Supplement: Combination bilberry/oats — The dietary intervention will be continued for three months. After randomization, participants will be given bilberry shakes (active), liquid oat shakes (active), a combination shake with bilberry and oats, or reference shakes (placebo product containing no active bilberry or active oats but with similar taste and texture), for intake two times a day (t.i.d). The formula for the shakes to be used in the intervention will be finalized during the initial project period.
  Arms: Combination of oat and bilberry

SUMMARY:
Background:

Bilberries from Sweden, rich in polyphenols, have shown cholesterol-lowering effects in small studies, and the cholesterol-lowering properties of oats, with abundant beta-glucans and potentially bioactive phytochemicals, are well established. Both may provide cardiometabolic benefits for patients with manifest chronic cardiometabolic disease, such as type 2 diabets mellitus (T2DM) and myocardial infarction (MI). However, large studies of adequate statistical power and appropriate duration are needed to confirm clinically relevant treatment effects. No previous study has evaluated the potential additive or synergistic effects of bilberry combined with oats on cardiometabolic risk factors.

Design:

This is a double-blind, randomized, placebo-controlled clinical trial. Our primary objective is to assess cardioprotective effects of diet supplementation with dried bilberry and with bioprocessed oat bran, with a secondary explorative objective of assessing their combination, compared with a neutral isocaloric reference supplement, for patients diagnosed with T2DM and/or MI. Patients will be randomized 1:1:1:1 to a three-month intervention. The primary endpoint is the difference in LDL cholesterol change between the intervention groups after three months. The major secondary endpoint is exercise capacity at three months. Other secondary endpoints include plasma concentrations of biochemical markers of inflammation, glycaemia, and gut microbiota composition after three months.

Implications:

Secondary prevention after cardiometabolic disease, including T2DM and MI, has improved during the last decades but diabetes complications, readmissions and cadiovascular related deaths following these conditions remain large health care challenges. Controlling hyperlipidemia, hyperglycaemia, hypertension and inflammation is critical to preventing (new) cardiovascular events, but novel pharmacological treatments for these conditions are expensive and associated with negative side effects. If bilberry and/or oat, in addition to standard medical therapy, can lower LDL cholesterol and inflammation more than standard therapy alone, this could be a cost-effective and safe dietary strategy for secondary prevention in high-risk patients or risk prevention in subjects with T2DM.

ELIGIBILITY:
Inclusion criteria

* Confirmed T2DM diagnosis (any treatment modality accepted) and/or within 3 years post STEMI or NSTEMI
* Completed coronary angiography/PCI
* Male and female subjects ≥18 years
* Allocated to atorvastatin at a daily dose of 80 mg (only eligible for patients enrolled up to 7 days post MI and not for T2D subjects)
* Written informed consent

Exclusion criteria

* Emergency coronary artery bypass grafting
* <18 years of age
* LDL cholesterol <2.0 mmol/L
* Daily intake or the intent to initiate daily intake of bilberry in any form or daily intake of >15 g of oatmeal or equivalent
* Food allergy/intolerance to gluten, bilberries or legumes
* Previous randomization in the BioDiaMI trial
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma levels of LDL cholesterol | Three months
  The effect of intervention on difference between the groups of LDL cholesterol after three months

SECONDARY OUTCOMES:
Plasma lipid profile | Three months
  The effect of intervention on differences between the groups of fasting lipid profile including HDL, triglycerides, total cholesterol, small-dense LDL cholesterol, apo A, apo B, Lp(a) and oxidized LDL.
Symptom-limited bicycle ergometer test | Three months
  The effect of intervention on exercise capacity (measured as maximal workload in Watts and as estimated maximal oxygen uptake (VO2 max))
Dynamic unilateral heel-lft and unilateral shoulder flexion tests | Three months
  The effect of intervention on muscle endurance
Self-reported physical activity level | Three months
  The effect of intervention on the Frändin/Grimby activity scale (6 levels of physical activity, min:1 (low activity) max:6 (heavy activity)) and the Haskell physical activity scale ("For how many days were you physically active during the last week for at least 20 minutes?", min:0 max:7)
Plasma concentrations of inflammatory and heart function markers | Three months
  The effect of intervention on plasma concentrations of biochemical markers of troponin, NT-proBNP, hs_CRP (high sensitivity C-reactive protein), IL-6 and HbA1c (glycosylated hemoglobin).
Plasma concentrations of other biochemical markers | Three months
  The effect if intervention on plasma concentrations of biochemical markers of insulin, creatinine, Cystatin C, glucose and C-peptide
Untargeted plasma metabolome | Three months
  Untargeted plasma metabolomics will be employed to exploratively assess alterations in endogenous and exposome-related metabolites and to identify metabolites that may differ with treatment.
Fecal samples of gut microbiota composition | Three months
  These exploratory analyses of will allow to investigate the extent to which gut microbiota composition and activity differs between responders and non-responders to the interventions.
Left ventricular systolic function | Three months
  The effect of intervention on left ventricular function. Baseline left ventricular systolic function, expressed as global ejection fraction in percent according to the biplane Simpson method, will be evaluated by echocardiography by the discharging physician. The procedure will be repeated after three months by an experienced echocardiography technician blinded to results of the initial examinations
Resting heart rate | Three months
  The effect of intervention on resting heart rate
Systolic and diastolic blood pressure | Three months
  The effect of intervention on blood pressure (mmHg)
Urine albumin-creatinine ratio | Three months
  Urine albumin-creatinine ratio will be measured for for T2DM only
Continuous glucose monitoring with Continuous Glucose Monitors (CGM) - FreeStyle model 2 | Three months
  Continuous glucose monitoring (in a subset of T2DM only, n=80 in total)
Body composition with multi-frequency biothesiometry | Three months
  Body composition willbe measured with multi-frequency biothesiometry (for T2DM only)

CONTACTS AND LOCATIONS:
Overall Officials: Ole Frobert, Prof, Study Director — Department of Cardiology, Örebro Univerity Hospital, 701 85 Örebro, Sweden; Cecilia Bergh, PhD, Principal Investigator — Clinical Epidemiology and Biostatistics, School of medical Sciences, örebro University, Sweden
Locations (8):
- Denmark (2):
  - Steno Diabetes center, Aarhus
  - Odense University Hospital, Odense
- Sweden (6):
  - Falu lasarett, Falun
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Karlstad general hospital, Karlstad
  - Department of Cardiology, Skånes universitetssjukhus, Lund
  - Department of Cardiology, Örebro University Hospital, Örebro
  - Cardiology Clinic, Västmanlands sjukhus, Västerås

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bergh C, Landberg R, Andersson K, Heyman-Linden L, Rascon A, Magnuson A, Khalili P, Karegren A, Nilsson J, Pirazzi C, Erlinge D, Frobert O. Effects of Bilberry and Oat intake on lipids, inflammation and exercise capacity after Acute Myocardial Infarction (BIOAMI): study protocol for a randomized, double-blind, placebo-controlled trial. Trials. 2021 May 10;22(1):338. doi: 10.1186/s13063-021-05287-5. PMID 33971938